CLINICAL TRIAL: NCT06666023
Title: The Diagnostic Pillar for Diagnosis of Infections in the Orthopedic Field: Smart and Sustainable Paper-based Electrochemical Point-of-care Device Assisted by Artificial Intelligence
Brief Title: Paper-based Electrochemical Point-of-care Device in Diagnostic of Orthopedic Infections
Acronym: Ortho-PoC
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Ministero della Salute, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: PNRR-POC-2023-12378291
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-09

CONDITIONS: PJI; Spondylodiscitis
Keywords: infections;; orthopedic surgery;; sensor;; PJI,; spondylodiscitis
MeSH Terms: conditions — Discitis; Infections | interventions — Equipment and Supplies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infection Group: Patients affected by PJI and Spondylodiscitis
  Interventions: Device: Device
- Control Group: Patients with post-contusive or inflammatory or arthritic suffusion
  Interventions: Device: Device

INTERVENTIONS:
Device: Device — Use of the device in groups to test its ability to diagnose infections.

SUMMARY:
Periprosthetic Joint infections (PJI) and spondylodiscitis are considered some of the most costly infectious diseases because require at least one surgery, prolonged hospitalisation, rehabilitation care, prolonged antibiotherapy, and extended absence from work in working-age patients. Ortho-PoC will face this issue with a smart and highly innovative diagnostic tool, starting from the point-of-care device for infection diagnosis in the orthopedic field developed and published by the coordinator Fondazione Policlinico Universitario Agostino Gemelli IRCCS and one partner Università degli Studi di Roma Tor Vergata. Ortho-PoC will further go beyond the state of the art by delivering a point-of-care device based on multiparametric analysis, in easily collected synovial fluids or pus. Several samples will be analysed using Ortho-PoC at three different Hospitals (Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Ospedali Riuniti di Foggia, Azienza Ospedaliera Universitaria Policlinico Vanvitelli Napoli) and the data will be treated with artificial intelligence (AI) to deliver an AI-assisted robust, effective, and smart diagnostic device for PJI.

ELIGIBILITY:
Inclusion Criteria:

* patients that received a joint implant or spine surgery, clear signs of infection (according to international guidelines)
* patients off antibiotic therapy at least for two weeks
* Sample biopsy of minimum 1 ml.

Exclusion Criteria:

* pregnant women,
* patient affected by cancer
* patient under antibiotic therapy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with a suspected history of PJI or spondylodiscitis according to international guidelines and subsequent diagnostic confirmation of infection.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity | at enrollement
  Most reliable cut-off evaluation in terms of best sensitivity and specificity of device in diagnosing PJI and spondylodiscitis

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Maccauro, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Rome, Lazio, Italy